CLINICAL TRIAL: NCT06770556
Title: An Investigation of TMS Effects Using Magnetoencephalography (MEG) Among Individuals With and Without Heavy Alcohol Use
Brief Title: Transcranial Magnetic Stimulation (TMS) Effects Using Magnetoencephalography (MEG) Study
Acronym: TMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00123420
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence; Alcohol Consumption
Keywords: Transcranial Magnetic Stimulation (TMS); Magnetoencephalography (MEG); Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Four Day - Option 1 (Other): Participants will receive active iTBS, sham iTBS, 10 Hz, 1 Hz.
  Interventions: Device: Sham iTBS; Device: Active iTBS; Device: 10 Hz TMS; Device: 1 Hz TMS
- Two Day - Option 1 (Other): Participants will receive active iTBS then sham iTBS.
  Interventions: Device: Sham iTBS; Device: Active iTBS
- Four Day - Option 2 (Other): Participants will receive sham iTBS, active iTBS, 1 Hz, 10 Hz.
  Interventions: Device: Sham iTBS; Device: Active iTBS; Device: 10 Hz TMS; Device: 1 Hz TMS
- Two Day - Option 2 (Other): Participants will receive sham iTBS then active iTBS.
  Interventions: Device: Sham iTBS; Device: Active iTBS

INTERVENTIONS:
Device: Sham iTBS — Participants will receive sham iTBS
Device: Active iTBS — Participants will receive active iTBS
Device: 10 Hz TMS — Participant will receive 10 Hz TMS
  Arms: Four Day - Option 1; Four Day - Option 2
Device: 1 Hz TMS — Participant will receive 1 Hz TMS
  Arms: Four Day - Option 1; Four Day - Option 2

SUMMARY:
Alcohol use disorder (AUD) is a complex chronic brain disease characterized by compulsive alcohol use, loss of control over drinking, and negative emotional states. Extensive research has identified the general neural circuitry underlying AUD. There is an exciting opportunity to intervene in AUD using neuromodulation. Transcranial magnetic stimulation (TMS) offers a non-invasive method to modulate brain activity, making it a promising tool for investigating, modulating, and potentially treating AUD. However, the precise effects of TMS on neural circuits involved in AUD and the mechanisms underlying these effects must first be understood. Magnetoencephalography (MEG) is a neuroimaging method that provides direct measurement of brain activity within neural circuits with high temporal resolution. Critically, MEG can measure brain activity in a wide range of frequencies that are consistent with those targeted by TMS. The goal of this proposal is therefore to collect preliminary and feasibility data to support a future NIH grant application that would use MEG to investigate TMS effects in individuals with AUD (iAUD).

DETAILED DESCRIPTION:
This proposal uses a mixed, between-group, within-subject design. The study will investigate the acute effects of different TMS pulse sequences in participants without AUD (non-AUD), and compare active/sham iTBS across non-AUD and AUD. On each study day, participants will complete a pre-TMS baseline MEG scan (10 min resting state), followed by a TMS pulse sequence, then complete 3 more MEG scans (immediately post-TMS, 1 hour post-TMS, and 2 hours post-TMS). Each TMS pulse sequence will be administered on a separate day and will be matched by the number of pulses administered (1200 pulses) and the total duration of administration time (20 min). The sham condition will control for auditory and sensory side effects associated with TMS. TMS will be applied to the left DLPFC, identified by the EEG F3 coordinate. Participants will either complete 4 study visits (n = 5) and receive 1 Hz, 10 Hz, iTBS, and sham, each on a separate day; or participants will complete 2 study visits (n = 5) and receive iTBS and sham, each on a separate day. Participants will also receive a structural MRI scan in order to map the MEG outcome data onto their own anatomical brain image.

ELIGIBILITY:
Inclusion Criteria non-AUD Participants:

* Diagnostic and Statistical Manual of Mental Disorders (DSM-5) score for AUD = 0
* Alcohol Use Disorders Identification Test (AUDIT) score ≤ 7
* Is not a heavy alcohol consumer

Inclusion Criteria AUD Participants:

* DSM-5 score for AUD ≥ 3
* AUDIT score ≥ 8
* Is a heavy alcohol consumer

Exclusion Criteria:

* Current substance use disorder other than alcohol use disorder and/or frequent use of non-prescribed psychoactive substances.
* Current serious psychiatric disorder, and/or any history of a psychotic disorder
* Any health problem that would interfere with the study or could be aggravated by study procedures (e.g., history of migraines, claustrophobia).
* Is currently taking or initiates a medication known to affect alcohol intake and/or craving.
* History of traumatic brain injury resulting in hospitalization, loss of consciousness, and/or having ever been informed he/she has an epidural, subdural, or subarachnoid hemorrhage.
* Does not meet safety criteria for TMS or MRI.
* Females of childbearing potential who are pregnant (by urine HCG), planning to become pregnant, nursing, or who are not using a reliable form of birth control.
* Is at an elevated risk of seizure (i.e. has a history of seizures, is currently prescribed medications known to lower seizure threshold and has had a change in their medication).
* Clinical Intake Withdrawal Assessment (CIWA>5) (to prevent delivering TMS to individuals in withdrawal).
* Not able to read and understand questionnaires, assessments, and/or the informed consent.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events Potentially Related to TMS | Through study completion 1 year
  The number of potential adverse events queried after each TMS session.

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No